CLINICAL TRIAL: NCT04935892
Title: Impact of Wearing Slippers on Transfer of Bacteriophage MS2 From Floors in Patient Rooms to Bedding and Surfaces
Brief Title: Slippers to Reduce Transfer From Floors to Surfaces
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louis Stokes VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr. Curtis Donskey, Principal Investigator, Louis Stokes VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17044-H34
Record Dates: First submitted 2021-06-12; First posted 2021-06-23 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Transmission, Other/Miscellaneous
Keywords: Floor; Bacteriophage MS2; Contamination; Environment; Healthcare-associated pathogens

STUDY DESIGN:
Intervention Model Description: Randomized trial
Who Masked: Outcomes Assessor
Masking Description: Lab personnel processing cultures blinded to the study group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Slippers (Experimental): Patients wear slippers any time they are out of bed with a goal of avoiding any contact between socks/feet and the floor
  Interventions: Behavioral: Slippers
- Control (No Intervention): Patients receive standard care with no intervention

INTERVENTIONS:
Behavioral: Slippers — Patients in the intervention group wear slippers when out of bed
  Arms: Slippers

SUMMARY:
The goal of this study is to determine if wearing slippers will reduce transfer of bacteriophage MS2 from hospital room floors to surfaces in the room and hands of patients. Subjects are randomized to wear slippers versus standard care and cultures are collected at 24 and 48 hours to assess transfer of bacteriophage MS2 from the floor to high-touch surfaces, personal items, bedding, socks or feet, and hands of patients.

DETAILED DESCRIPTION:
The goal of this study is to determine if wearing slippers will reduce transfer of bacteriophage MS2 from hospital room floors to surfaces in the room and hands of patients. Hospitalized patients are enrolled and randomized to wear slippers any time they are out of bed versus standard care. Bacteriophage MS2 is inoculated onto a site on the floor between the patient bed and the bathroom. Cultures are collected at 24 and 48 hours to assess transfer of bacteriophage MS2 from the floor to high-touch surfaces (bed rail, bedside table, telephone, call button), personal items, bedding, socks or feet, and hands of patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of 18 years of age or older
* Ambulatory
* Able to demonstrate an understanding of study procedures

Exclusion Criteria:

* Unable or unwilling to fulfill study requirements.
* Expected length of stay less than 48 hours
* Any patient deemed not suitable for study participation at the discretion of the study investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Contamination of a composite of high-touch surfaces, personal items, socks/feet, bedding, and hands | 48 hours
  Cultures for MS2

CONTACTS AND LOCATIONS:
Overall Officials: Curtis J Donskey, MD, Principal Investigator — Cleveland VA Medical Center
Locations (1):
- Cleveland VA Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
We will provide de-identified individual participant data to those who provide a request in writing.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Available 6/22/21 through 6/22/24
Access Criteria: Written request

REFERENCES:
- [Derived] Haq MF, Alhmidi H, Redmond SN, Cadnum JL, Silva SY, Wilson BM, Donskey CJ. A randomized trial to determine whether wearing slippers reduces transfer of bacteriophage MS2 from floors to patients and surfaces in hospital rooms. Infect Control Hosp Epidemiol. 2023 Apr;44(4):670-673. doi: 10.1017/ice.2021.475. Epub 2022 Aug 23. PMID 35997135

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT04935892/SAP_000.pdf